CLINICAL TRIAL: NCT05118750
Title: An Open-label Study of ALTO-300 in Adults With Major Depressive Disorder
Brief Title: ALTO-300 in Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alto Neuroscience (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTO-300-002
Record Dates: First submitted 2021-10-18; First posted 2021-11-12 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALTO-300 (Experimental): ALTO-300 oral (PO) tablet; daily dosing 8 weeks
  Interventions: Drug: ALTO-300 oral (PO) tablet

INTERVENTIONS:
Drug: ALTO-300 oral (PO) tablet — One tablet daily

SUMMARY:
The purpose of this study is to collect biologically-based data for defining predictors and correlates of the effects of ALTO-300.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of MDD based on the Structured Clinical Interview for DSM-5 (SCID) for depression
* have moderate to severe depression on DSM-5 depression criteria items, as assessed by a score of ≥10 on the Patient Health Questionnaire-9 (PHQ-9) at each of Visits 1, 2, and 3
* at baseline (Visit 2) are taking a stable dose of a single SSRI, serotonin-norepinephrine reuptake inhibitor (SNRI), or bupropion and have been on that medication for ≥6 weeks at an adequate dosage defined by the Antidepressant Treatment Response Questionnaire (ATRQ), and with no modification to dosage for ≥2 weeks.
* have either: had a continuous period of euthymia of at least 2 months in the past 26 months, regardless of the number of failed antidepressants OR not had a period of euthymia of at least 2 months in the past 26 months but within the past 24 months have not failed >3 antidepressants at an adequate dosage and duration as defined by the ATRQ
* are currently on their last failed currently prescribed permitted baseline antidepressant medication
* have a response to their currently prescribed antidepressant noted as depression that has improved ≤49% as defined by the ATRQ.
* agree to, and are eligible for all biomarker assessments (EEG, neurocognitive testing, activity and sleep monitoring, genetic testing). To participate in the activity and sleep monitoring biomarkers, all participants will be required to have a smart phone or an internet enabled tablet. A participant who otherwise qualifies may refuse the salivary genetic sample and be included in the study.
* fluent in English
* willing to comply with all study procedures (with the notes above), able to complete all assessments independently, and available for the duration of the study.

Exclusion Criteria:

Any of the following medical conditions:

* hepatic impairment (i.e., cirrhosis or active/chronic liver disease)
* baseline serum transaminase levels that exceed 2x upper limit of normal(ULN)
* severe impediment to vision, hearing, comprehension, and/or hand movement that interferes with study tasks.
* any contraindications to EEG (i.e., requiring high concentration oxygen)
* active suicidal ideation as assessed by the investigator.
* moderate to severe Alcohol Use Disorder (AUD)

Concurrent use of any of the following at baseline (Visit 2):

* tricyclic antidepressants (TCAs), mirtazapine, or monoamine oxidase inhibitors (MAOIs)
* melatonin, ramelteon, or other melatonin agonist
* a potent CYP1A2 inhibitor (e.g., fluvoxamine and ciprofloxacin)
* antipsychotics or mood stabilizers
* hypnotics, anxiolytics, stimulants, or opiate pain medications greater than three days per week and unable to reduce use to 3 or fewer days per week on an as needed basis

Have received electroconvulsive therapy (ECT), deep brain stimulation (DBS),vagus nerve stimulation (VNS), >2 treatments with ketamine, or esketamine in thecurrent depressive episode.

Diagnosis of bipolar disorder or a psychotic disorder based on the SCID forDSM-5

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
To understand the relationship between baseline biology and clinical outcome to ALTO-300 using the Montgomery-Åsberg Depression Rating Scale (MADRS) | Measured 6 times over 8 weeks
  The Montgomery-Åsberg Depression Rating Scale (MADRS) measures the severity of depression where smaller scores indicate less depression and higher scores suggest more severe depression. Possible scores for this 10 item version range from 0 to 60. The change from baseline to the end of the study is the primary outcome.
To understand the relationship between baseline biology and clinical outcome to ALTO-300 using the Clinical Global Impression scale - Severity (CGI-S) | Measured 6 times over 8 weeks
  The Clinical Global Impression scale - Severity (CGI-S) measures the severity of psychopathology in general where smaller scores indicate less illness and higher scores suggest more severe illness. Possible scores for this scale range from 1 to 7. The change from baseline to the end of the study is the primary outcome.
To evaluate the safety of ALTO-300 | From the signing of the ICF until the follow-up visit (up to 12 weeks)
  Incidence, severity, and relatedness of TEAEs,SAEs, discontinuation due to TEAEs, and deaths
To evaluate the safety of ALTO-300 | From the signing of the ICF until the end-of-treatment visit (up to 11 weeks)
  Assessment of vital signs and laboratory data, withparticular attention to liver function tests

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Site 153, Culver City, California
  - Site 103, Sacramento, California
  - Site 158, Santee, California
  - Site 159, Clermont, Florida
  - Site 161, Okeechobee, Florida
  - Site 137, Noblesville, Indiana
  - Site 166, Saint Charles, Missouri
  - Site 132, New York, New York
  - Site 102, Dallas, Texas
  - Site 165, DeSoto, Texas
  - Site 147, Fort Worth, Texas